CLINICAL TRIAL: NCT05407259
Title: Investigating the Inverted-U Relationship Between Cognitive Performance and Plasma Epinephrine: A Registered Report of a Four-arm Crossover Randomized Controlled Trial
Brief Title: Investigating the Inverted-U Relationship Between Cognitive Performance and Plasma Epinephrine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Ting-Yu Lin, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202205HM003
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Healthy Young Adults
Keywords: Resistance Training; Kinesiology, Applied; Cognitive Neuroscience; Psychology, Sports; Cognitive Psychology; Psychophysiology; Exercise; Circuit-Based Exercise
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Masking Description: Blinding (masking) and controlling risk of bias Because of the nature of exercise interventions, the blinding of participants and experimenters is not applicable to our study. To reduce the threat of the placebo effect, we will ask participants for their expectations on cognitive performance, and these will be incorporated into our statistical analysis. Blinding of the outcome assessors is also not possible. However, all measurements of cognitive performance will be computerized and not involve human judgment. The data analyzers will not be blinded but will follow a pre-specified statistical analysis plan. These procedures will reduce the risk of bias arising from the lack of blinding of participants, experimenters, assessors, and data analyzers and the threat from researchers' degrees of freedom.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control condition (No Intervention): During the control condition, participants will be asked to read a book related to exercise for approximately 40 minutes.
- Low-intensity barbell resistance exercise (Experimental): Exercise: Barbell squat, barbell press, and barbell deadlift Number of sets: 3 Number of repetitions: 5 Intensity: 65% 1RM Training method: Circuit training (Squat set 1 ➔ Press set 1 ➔ Deadlift set 1 ➔ Squat set 2 ➔ Press set 2 ➔ Deadlift set 2 ➔ Squat set 3 ➔ Press set 3 ➔ Deadlift set 3) Rest interval between exercises and sets: ~3 minutes (Warm-up: 1 set of 5 repetitions for each exercise at 50% 1RM)
  Interventions: Behavioral: Resistance exercise
- Moderate-intensity barbell resistance exercise (Experimental): Exercise: Barbell squat, barbell press, and barbell deadlift Number of sets: 3 Number of repetitions: 5 Intensity: 72% 1RM Training method: Circuit training (Squat set 1 ➔ Press set 1 ➔ Deadlift set 1 ➔ Squat set 2 ➔ Press set 2 ➔ Deadlift set 2 ➔ Squat set 3 ➔ Press set 3 ➔ Deadlift set 3) Rest interval between exercises and sets: ~3 minutes (Warm-up: 1 set of 5 repetitions for each exercise at 50% 1RM)
  Interventions: Behavioral: Resistance exercise
- High-intensity barbell resistance exercise (Experimental): Exercise: Barbell squat, barbell press, and barbell deadlift Number of sets: 3 Number of repetitions: 5 Intensity: 78% 1RM Training method: Circuit training (Squat set 1 ➔ Press set 1 ➔ Deadlift set 1 ➔ Squat set 2 ➔ Press set 2 ➔ Deadlift set 2 ➔ Squat set 3 ➔ Press set 3 ➔ Deadlift set 3) Rest interval between exercises and sets: ~3 minutes (Warm-up: 1 set of 5 repetitions for each exercise at 50% 1RM)
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Resistance exercise — There will be four conditions (three exercises and one control) on visits 3-6. For the three exercise conditions, all training parameters except intensity will be the same. The sets in high, moderate, and low intensity correspond to the rate of perceived exertion (0-10 scale) 7-9, 5-6, and 3-4, respectively. Therefore, the participants will perform 5 repetitions barbell squat, barbell press, and barbell deadlift with 8RM (78% 1RM), 11RM (72% 1RM), and 16RM (65% 1RM) for 3 sets
  Other Names: Resistance training
  Arms: High-intensity barbell resistance exercise; Low-intensity barbell resistance exercise; Moderate-intensity barbell resistance exercise

SUMMARY:
Abstract Although acute resistance exercise has been suggested to enhance inhibitory control, a critical component of executive function, the mechanism by which acute exercise influences inhibitory control is unclear and there are methodological limitations in previous empirical studies. According to the locus coeruleus-norepinephrine (LC-NE) theory, the activity of the LC, the major releaser of NE in the brain, regulates inhibitory control. Because there is reciprocal communication between circulating epinephrine and the LC. Plasma epinephrine is chosen as the index of LC-NE activity. However, only one study in acute exercise-inhibitory control measured the plasma epinephrine. Therefore, this registered report aims to extend its findings by a four-arm crossover randomized controlled design with three different intensities, using free-weight, multiple-joint, and structural resistance exercises. Moreover, most studies showed some methodological limitations such as failing to report the process of randomization, implementing a familiarization of resistance exercise before the maximal strength test, and publishing the protocol. Without a transparent report on how the participants were allocated, the results were at risk of bias. Without a familiarization of resistance exercise, the maximal muscle strength was likely to be underestimated. Without publishing the protocol before data collection, these findings were threatened by undetected researchers' degrees of freedom such as HARKing (hypothesizing after the results are known), cherry picking, and p-hacking. This registered report will address the limitations of previous studies by incorporating cognitive and resistance exercise familiarization, transparently reporting the randomization process, and submitting it as a registered report.

ELIGIBILITY:
Inclusion Criteria:

1. healthy young male aged 18-40 years;
2. recreational resistance-trained (≥ 1 time/week for the previous 6 months);
3. free from cardiovascular, cerebrovascular, and neurological disorders and other chronic diseases;
4. free from any medical condition listed on the 2014 update of the Physical Activity Readiness Questionnaire (PAR-Q+);
5. non-smoker; and
6. normal or corrected-to-normal vision.

Exclusion Criteria:

1. athlete trained in a competitive sports team or engaging in exercise for more than 20 hours/week;
2. unable to perform any of the intervention exercises (barbell squat, press, and deadlift); or
3. color blind

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Inhibitory control (change between baseline and 5 minutes after intervention/control) | Baseline (before intervention) and 5 minutes after (post-task) intervention/control.
  The Inhibitory control (Stroop interference score) will be the mean incongruent reaction time minus the mean congruent reaction time. Lower scores mean a better outcome.
Inhibitory control (change between baseline and 20 minutes after intervention/control) | Baseline (before intervention) and 20 minutes after (post-task) intervention/control.
  The Inhibitory control (Stroop interference score) will be the mean incongruent reaction time minus the mean congruent reaction time. Lower scores mean a better outcome.
Inhibitory control (change between baseline and 35 minutes after intervention/control) | Baseline (before intervention) and 35 minutes after (post-task) intervention/control.
  The Inhibitory control (Stroop interference score) will be the mean incongruent reaction time minus the mean congruent reaction time. Lower scores mean a better outcome.
Inhibitory control (change between baseline and 50 minutes after intervention/control) | Baseline (before intervention) and 50 minutes after (post-task) intervention/control.
  The Inhibitory control (Stroop interference score) will be the mean incongruent reaction time minus the mean congruent reaction time. Lower scores mean a better outcome.
Information processing speed (change between baseline and 5 minutes after intervention/control) | Baseline (before intervention) and 5 minutes after intervention/control.
  The Information processing speed will be the mean simple reaction time. Lower scores mean a better outcome.
Information processing speed (change between baseline and 20 minutes after intervention/control) | Baseline (before intervention) and 20 minutes after intervention/control.
  The Information processing speed will be the mean simple reaction time. Lower scores mean a better outcome.
Information processing speed (change between baseline and 35 minutes after intervention/control) | Baseline (before intervention) and 35 minutes after intervention/control.
  The Information processing speed will be the mean simple reaction time. Lower scores mean a better outcome.
Information processing speed (change between baseline and 50 minutes after intervention/control) | Baseline (before intervention) and 50 minutes after intervention/control.
  The Information processing speed will be the mean simple reaction time. Lower scores mean a better outcome.

SECONDARY OUTCOMES:
Epinephrine (change between baseline and immediately after intervention/control) | Baseline and immediately after intervention/control.
  Plasma epinephrine concentrations will be measured in duplicate using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Epinephrine (change between baseline and 15 minutes after intervention/control) | Baseline and 15 minutes after intervention/control.
  Plasma epinephrine concentrations will be measured in duplicate using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Epinephrine (change between baseline and 30 minutes after intervention/control) | Baseline and 30 minutes after intervention/control.
  Plasma epinephrine concentrations will be measured in duplicate using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Epinephrine (change between baseline and 45 minutes after intervention/control) | Baseline and 45 minutes after intervention/control.
  Plasma epinephrine concentrations will be measured in duplicate using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Epinephrine (change between baseline and 60 minutes after intervention/control) | Baseline and 60 minutes after intervention/control.
  Plasma epinephrine concentrations will be measured in duplicate using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.

IPD SHARING:
Plan to Share IPD: Yes
We will publish the raw data online when we submit the resulting manuscript.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol is available on Open Science Framework (https://osf.io/4fkpc/).
  The raw data will be published after the trial is completed. (No time limitation imposed)
Access Criteria: No limitation.
URL: https://osf.io/4fkpc/

REFERENCES:
- See also: Related Info — https://osf.io/4fkpc/